CLINICAL TRIAL: NCT01953367
Title: Bioequivalence and Safety Study of Vantobra and TOBI Nebulizer Solutions in Healthy Subjects
Brief Title: Bioequivalence and Safety of Vantobra and TOBI in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12012.102
Record Dates: First submitted 2013-09-04; First posted 2013-10-01 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Cystic Fibrosis
Keywords: Bioequivalence; AUC; Cmax
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vantobra; Treatment A (Experimental): Vantobra, 170 mg tobramycin/1.7 mL nebulizer solution
  Interventions: Drug: Vantobra (tobramycin)
- TOBI; Treatment B (Active Comparator): TOBI, 300 mg tobramycin/5 mL nebulizer solution
  Interventions: Drug: TOBI (tobramycin)

INTERVENTIONS:
Drug: Vantobra (tobramycin) — Inhalation
  Arms: Vantobra; Treatment A
Drug: TOBI (tobramycin) — Inhalation
  Arms: TOBI; Treatment B

SUMMARY:
This study will investigate the bioequivalence and compare the safety profiles following inhalation of Vantobra to TOBI nebulizer solution in healthy subjects.

Bioequivalence will be investigated based on the pharmacokinetic plasma profiles of Vantobra nebulizer solution compared to TOBI nebulizer solution.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects of any ethnic origin
* Aged between 18 and 50 years of age
* Body weight of ≥50 kg and body mass index (BMI) between 18.5 and 29 kg/m2
* FEV1 > 90% of predicted
* Able to demonstrate correct inhaler use
* Written informed consent

Exclusion Criteria:

* History of clinically relevant allergies or idiosyncrasies to tobramycin or any other inactive ingredient(s) of the IMP
* Any history of drug hypersensitivity, asthma, urticaria, or other significant allergic diathesis.
* Any evidence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinological, metabolic, neurological, psychiatric or other diseases at screening
* Surgery of the gastrointestinal or respiratory tract which might interfere with drug absorption
* History of malignancy within the past 5 years
* History of orthostatic hypotension, faintings or blackouts
* Acute or chronic viral, bacterial or fungal airway infections, including laryngeal infections, mouth and throat infections, and hoarseness;
* Other clinically relevant chronic or acute infectious illnesses
* Clinical chemical, hematological or any other laboratory parameters clinically relevant outside the normal range

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To investigate the bioequivalence (in terms of relative systemic bioavailability based on pharmacokinetic plasma profiles) of Vantobra 170 mg/1.7 mL nebulizer solution as compared to TOBI 300 mg/5 mL nebulizer solution in healthy subjects | Day 1 and Day 7
  Plasma AUClast of tobramycin
To investigate the bioequivalence (in terms of relative systemic bioavailability based on pharmacokinetic plasma profiles) of Vantobra 170 mg/1.7 mL nebulizer solution as compared to TOBI 300 mg/5 mL nebulizer solution in healthy subjects | Day 1 and Day 7
  Plasma Cmax of tobramycin
To investigate the bioequivalence (in terms of relative systemic bioavailability based on pharmacokinetic plasma profiles) of Vantobra 170 mg/1.7 mL nebulizer solution as compared to TOBI 300 mg/5 mL nebulizer solution in healthy subjects | Day 1 and Day 7
  tmax of tobramycin

SECONDARY OUTCOMES:
Number of Adverse Events during the trial period | Adverse Events during the study period of max. 17 days
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wolgang Timmer, MD, Principal Investigator — Inamed GmbH
Locations (1):
- Inamed GmbH, Gauting, Germany